CLINICAL TRIAL: NCT02876588
Title: Assessing the Risk of Wrong-Patient Errors in an Electronic Health Record That Allows Multiple Records Open
Brief Title: Risk of Wrong-Patient Errors With Multiple Records Open
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAQ9954; R21HS023704 (AHRQ)
Record Dates: First submitted 2016-08-03; First posted 2016-08-24 (Estimated); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Medical Errors; Medical Order Entry Systems
Keywords: Wrong-Patient Errors; Retract-and-Reorder measure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unrestricted (Active Comparator): Users have "unrestricted" access to open up to a maximum of 4 patient records at a time in the EHR
  Interventions: Other: Unrestricted
- Restricted (Active Comparator): Users have "restricted" access to open a maximum of 1 patient record at a time in the EHR
  Interventions: Other: Restricted

INTERVENTIONS:
Other: Unrestricted — Users may open up to 4 patient records at a time.
  Arms: Unrestricted
Other: Restricted — Users are restricted to open 1 patient record at a time.
  Arms: Restricted

SUMMARY:
This study is designed to achieve the following aims:

1. Assess the relationship between the number of records open at the time of placing an order, and the risk of placing an order on the wrong patient.
2. Compare the incidence of wrong-patient orders in a "restricted environment" that limits its providers to only one record open at a time to an "unrestricted environment" where users can open a maximum of four records at once.
3. The results of this study will help inform decisions on how to safely implement EHR systems.
4. The results of this study will inform a larger scale health IT implementation research project evaluating the balance between the wrong-patient error risks and potential efficiency gains of having multiple records open at once, with rigorous research methodologies.

DETAILED DESCRIPTION:
Currently, at least 70,000 U.S. physicians use computerized provider order entry (CPOE) to place orders. This number is expected to rise sharply as hospitals continue to take advantage of federal incentives and adopt electronic health record (EHR) technology. Although CPOE is associated with a reduction in medical errors, when orders are placed electronically certain types of errors, including placing orders on the wrong patient, may occur more frequently.

Although there have been no studies quantifying (or even establishing) an increased risk of wrong-patient errors when providers have multiple records open at once, there have been several articles and expert opinions that warn of this potential risk.

The mechanism by which multiple patient records opened simultaneously can lead to a wrong-patient error may be related to the ease with which users can toggle between patient records and the similar looking computer screens. The magnitude of this risk needs to be established to help Information Technology (IT) leadership decide on how to safely implement CPOE systems.

There have been no studies demonstrating whether multiple records increase the risk of wrong-patient errors, by how much, and if any increase is dependent on the number of records open. This research project is an important first step in quantifying this risk.

In a randomized controlled trial conducted at Montefiore Medical Center, investigators propose to randomize inpatient and outpatient providers to a maximum of one record open at the time of ordering (restricted mode) or a maximum of four records open at the time of ordering (unrestricted mode).

Assignments will be made prior to the start of the study, and will remain constant throughout the study. A computer programmer working in IT, who is not an investigator of this study, will use Microsoft Excel to generate random numbers and assign one number to each provider. Providers assigned odd numbers will be in the restricted cohort, and those assigned even numbers will be in the unrestricted cohort. Providers who join Montefiore after the start of the study will be assigned a random number from Excel when assigned a new user log in for the EHR from a computer programmer not affiliated with the study, and will be added to the appropriate group based on their assigned random number. At the start of the randomized controlled trial, investigators will explain the purpose of the study to clinical staff via email and directly from within their IT systems, using a message crafted by the study team. The message will assure clinicians that data will be kept confidential and cooperation will carry no risk to them.

Montefiore uses the Epic Systems Corporation, or Epic, EHR system. Epic will implement the Retract-and-Reorder (RAR) tool, an automated method for identifying wrong-patient electronic orders, as well as capture the number of records open at the time of placing an order. This study will examine the effect of having the EHR system in restricted mode vs. unrestricted mode on RAR events. The goal is to obtain an estimate of the effect size and the intra-class correlations to provide preliminary data for a larger-scale health IT implementation research project. The unit of analysis will be the order. First, the RAR event rate for orders placed in the restricted vs. unrestricted mode will be calculated, testing the difference in rates using rank sum tests. Next, the relationship between the RAR event rate in restricted vs. unrestricted mode in subsets of providers and settings will be examined to determine whether specific types of providers or settings carry increased risk. Finally, a mixed-effects logistic regression model will be fitted with RAR event as the outcome and mode of the EHR system (restricted vs. unrestricted) as the independent variable of interest. The model will include random effects at the provider and order-session level because previous work has suggested substantial within-provider and within-session correlation. Orders will be nested in sessions and sessions will be nested in providers. To address the threat of confounding, the model will include fixed-effects variables including provider, patient, order-session, and order level covariates.

To safeguard against the possibility that the intervention actually worsens (increases) the RAR event rate, and to prevent unnecessary continuation of a study that is already conclusive, a data safety monitoring committee will conduct one interim review of the data in the randomized controlled trial.

ELIGIBILITY:
Clinician Participant Inclusion Criteria:

-All clinicians (physicians, nurse practitioners, physician assistants) who placed electronic orders during the study period will be included in the study. (Randomization is at the level of the clinician.)

Clinician Exclusion Criteria:

- Clinicians whose workflow requires access to more than one patient record at a time.

Patient Record Inclusion Criteria:

-All inpatient, emergency department, and ambulatory patients for whom electronic orders were placed during the study period will be included in the study.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3356 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Adelman, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Research may request data from the PI (Jason Adelman). Partial, de-identified order data will be made available for research purposes for analyses approved by the researchers' Institutional Review Board and by the PI. Data will be made available upon approval.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication of results.
Access Criteria: 1. Approval by the researchers' Institutional Review Board.
  2. Approval by the PI.

REFERENCES:
- [Background] Adelman J, Aschner J, Schechter C, Angert R, Weiss J, Rai A, Berger M, Reissman S, Parakkattu V, Chacko B, Racine A, Southern W. Use of Temporary Names for Newborns and Associated Risks. Pediatrics. 2015 Aug;136(2):327-33. doi: 10.1542/peds.2015-0007. Epub 2015 Jul 13. PMID 26169429
- [Background] Adelman JS, Kalkut GE, Schechter CB, Weiss JM, Berger MA, Reissman SH, Cohen HW, Lorenzen SJ, Burack DA, Southern WN. Understanding and preventing wrong-patient electronic orders: a randomized controlled trial. J Am Med Inform Assoc. 2013 Mar-Apr;20(2):305-10. doi: 10.1136/amiajnl-2012-001055. Epub 2012 Jun 29. PMID 22753810
- [Background] Adelman JS, Aschner JL, Schechter CB, Angert RM, Weiss JM, Rai A, Parakkattu V, Goffman D, Applebaum JR, Racine AD, Southern WN. Babyboy/Babygirl: A National Survey on the Use of Temporary, Nondistinct Naming Conventions for Newborns in Neonatal Intensive Care Units. Clin Pediatr (Phila). 2017 Oct;56(12):1157-1159. doi: 10.1177/0009922817701178. Epub 2017 Apr 12. No abstract available. PMID 28403654
- [Background] Adelman JS, Berger MA, Rai A, Galanter WL, Lambert BL, Schiff GD, Vawdrey DK, Green RA, Salmasian H, Koppel R, Schechter CB, Applebaum JR, Southern WN. A national survey assessing the number of records allowed open in electronic health records at hospitals and ambulatory sites. J Am Med Inform Assoc. 2017 Sep 1;24(5):992-995. doi: 10.1093/jamia/ocx034. PMID 28419267
- [Background] Adelman JS, Aschner JL, Schechter CB, Angert RM, Weiss JM, Rai A, Berger MA, Reissman SH, Yongue C, Chacko B, Dadlez NM, Applebaum JR, Racine AD, Southern WN. Evaluating Serial Strategies for Preventing Wrong-Patient Orders in the NICU. Pediatrics. 2017 May;139(5):e20162863. doi: 10.1542/peds.2016-2863. PMID 28557730
- [Background] Kannampallil TG, Manning JD, Chestek DW, Adelman J, Salmasian H, Lambert BL, Galanter WL. Effect of number of open charts on intercepted wrong-patient medication orders in an emergency department. J Am Med Inform Assoc. 2018 Jun 1;25(6):739-743. doi: 10.1093/jamia/ocx099. PMID 29025090
- [Background] Wachter RM, Murray SG, Adler-Milstein J. Restricting the Number of Open Patient Records in the Electronic Health Record: Is the Record Half Open or Half Closed? JAMA. 2019 May 14;321(18):1771-1773. doi: 10.1001/jama.2019.3835. No abstract available. PMID 31087007
- [Result] Adelman JS, Applebaum JR, Schechter CB, Berger MA, Reissman SH, Thota R, Racine AD, Vawdrey DK, Green RA, Salmasian H, Schiff GD, Wright A, Landman A, Bates DW, Koppel R, Galanter WL, Lambert BL, Paparella S, Southern WN. Effect of Restriction of the Number of Concurrently Open Records in an Electronic Health Record on Wrong-Patient Order Errors: A Randomized Clinical Trial. JAMA. 2019 May 14;321(18):1780-1787. doi: 10.1001/jama.2019.3698. PMID 31087021
- [Derived] Southern WN, Applebaum JR, Salmasian H, Kneifati-Hayek J, Carter EJ, Sumner JA, Adelman JS. Clinician Experience of Electronic Health Record Configurations Displaying 1 vs 4 Records at a Time. JAMA Intern Med. 2019 Dec 1;179(12):1723-1725. doi: 10.1001/jamainternmed.2019.3688. PMID 31524923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All clinicians who placed electronic orders during the study period at a large health system in New York in the emergency department (ED), inpatient, and outpatient settings.
Pre-assignment Details: Clinicians were excluded if their workflow included: 1) required 2 open patient records simultaneously (eg, mother-infant services), or 2) bypassed standard order entry process and could not be captured by the outcome measure (eg, radiologist).
Groups:
- Unrestricted: Users have "unrestricted" access to open a maximum of 4 patient records at a time in the Electronic Health Record (EHR)
Period: Overall Study
Arm/Group | Unrestricted | Restricted
Started | 1687 | 1669
Received Assigned Intervention | 1556 | 1400
Assigned to Opposite Group at Start of Trial Period (Assigned to opposite group at beginning of trial and remained in that group throughout the study.) | 120 | 185
Switched Groups During Trial Period (Switched groups during the trial and remained in that group for the duration of the study.) | 11 | 84
Completed (Observations (orders placed) for all randomized clinicians were included in the analysis. Assessments were performed according to randomized group (as randomized analysis) and per assignment received (as treated analysis).) | 1687 | 1669
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Clinicians with the authority to place an electronic order during the study period. Clinicians were excluded if their workflow included: 1) required 2 open patient records simultaneously (e.g., mother-infant services), or 2) bypassed standard order entry process and could not be captured by the outcome measure (e.g., radiologist).
Groups:
- Unrestricted: Users have "unrestricted" access to open a maximum of 4 patient records at a time in the EHR
- Total: Total of all reporting groups
Arm/Group | Unrestricted | Restricted | Total
Number analyzed (Participants) | 1687 | 1669 | 3356
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (12.3) | 42.9 (12.7) | 43.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 959 | 935 | 1894
  Male | 728 | 734 | 1462
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Experience at Study Site [Mean (Standard Deviation); unit: years] | 6.6 (6.0) | 6.4 (6.0) | 6.5 (6.0)
Provider Type [Count of Participants; unit: Participants]
  Attending Physician | 814 | 806 | 1620
  House staff | 542 | 529 | 1071
  Mid-level | 331 | 334 | 665

OUTCOME MEASURES:

1. Primary Outcome: Wrong-patient Order Sessions, Defined as Order Sessions That Include at Least One Wrong-Patient Retract-and-Reorder (RAR) Event, As-randomized Analysis
Description: The primary analysis included all order sessions performed by clinicians according to their assigned randomization group. The primary outcome was wrong-patient order sessions, defined as order sessions that include at least 1 wrong-patient Retract-and-Reorder (RAR) event.
  Wrong-patient order sessions were identified using the Wrong-Patient Retract-and-Reorder (RAR) measure. The Wrong-Patient RAR measure uses an electronic query to identify wrong-patient RAR events, defined as one or more orders placed for a patient that are retracted (cancelled) by the same provider within 10 minutes, and then reordered by the same provider for a different patient within the next 10 minutes.
Time Frame: 19-month study period. All order sessions placed by randomized clinicians during the study period were included in the analysis. The time frame for each participant varied.
Population: All clinicians with the authority to place an electronic order during the study period, grouped by their assigned randomization. Clinicians were excluded if their workflow: 1) required 2 open patient records simultaneously (eg, mother-infant services), or 2) bypassed standard order entry process and could not be captured by the outcome measure (eg, radiologist).
Measure: Number; unit: Wrong-patient order sessions
Units Other Than Participants: Order sessions
Arm/Group | Unrestricted | Restricted
Number analyzed (Participants) | 1687 | 1669
Number analyzed (Order sessions) | 6283306 | 5856992
Wrong-patient order sessions | 3015 | 3058
Statistical Analysis 1: Comparison: Unrestricted vs Restricted; Test type: Superiority; p = .60, Regression, Logistic — Random-effects logistic regression models were constructed, using RAR order sessions as the outcome, randomization group as the independent variable, and the clinician as the random intercept to account for nesting of order sessions within clinicians; Odds Ratio (OR) = 1.03, 95% CI 2-sided [.90 to 1.20]

2. Secondary Outcome: Wrong-patient Order Sessions, Defined as Order Sessions That Include at Least One Wrong-Patient Retract-and-Reorder (RAR) Event, as Treated Analysis
Description: The outcome was wrong-patient order sessions, defined as order sessions that include at least 1 wrong-patient Retract-and-Reorder (RAR) event. In the as treat analysis, each order was characterized by the clinician's initial configuration at the time an order was placed.
  Wrong-patient order sessions were identified using the Wrong-Patient Retract-and-Reorder (RAR) measure. The Wrong-Patient RAR measure uses an electronic query to identify wrong-patient RAR events, defined as one or more orders placed for a patient that are retracted (cancelled) by the same provider within 10 minutes, and then reordered by the same provider for a different patient within the next 10 minutes.
Time Frame: as for outcome 1
Population: Clinicians were grouped according to their configuration at the time an electronic order was placed. Clinicians were excluded if their workflow: 1) required 2 open patient records simultaneously (eg, mother-infant services), or 2) bypassed standard order entry process and could not be captured by the outcome measure (eg, radiologist).
Measure: Number; unit: Wrong-patient order sessions
Units Other Than Participants: Order sessions
Arm/Group | Unrestricted | Restricted
Number analyzed (Participants) | 1825 | 1531
Number analyzed (Order sessions) | 6415909 | 5724389
Wrong-patient order sessions | 3091 | 2982
Statistical Analysis 1: Comparison: Unrestricted vs Restricted; Test type: Superiority; p = .68, Regression, Logistic — Random-effects logistic regression models were constructed, using RAR order sessions as the outcome, randomization group as the independent variable, the clinician as the random intercept to account for nesting of order sessions within clinicians; Odds Ratio (OR) = 1.03, 95% CI 2-sided [.89 to 1.19]

3. Post Hoc Outcome: Wrong-patient Order Sessions, Defined as Order Sessions That Include at Least One Wrong-Patient Retract-and-Reorder (RAR) Event, Unrestricted Group
Description: The outcome measure was the rate of wrong-patient order sessions by the number of records open when orders were placed in the unrestricted group. Wrong-patient order sessions are defined as order sessions that include at least 1 wrong-patient Retract-and-Reorder (RAR) event.
  Wrong-patient order sessions were identified using the Wrong-Patient Retract-and-Reorder (RAR) measure. The Wrong-Patient RAR measure uses an electronic query to identify wrong-patient RAR events, defined as one or more orders placed for a patient that are retracted (cancelled) by the same provider within 10 minutes, and then reordered by the same provider for a different patient within the next 10 minutes.
  The outcome measure was reported as the number of wrong-patient order sessions per 100,000 order sessions.
Time Frame: as for outcome 1
Population: All clinicians with the authority to place an electronic order during the study period. Clinicians were excluded if their workflow included: 1) required 2 open patient records simultaneously (eg, mother-infant services), or 2) bypassed standard order entry process and could not be captured by the outcome measure (eg, radiologist).
Measure: Number; unit: wrong order sessions / 100,000 sessions
Units Other Than Participants: Order sessions
Groups:
- Unrestricted, 1 Record Open: Users have "unrestricted" access to open up to a maximum of 4 patient records at a time in the EHR
  Unrestricted, 1 record open: Users only opened 1 record at a time
- Unrestricted, 2 Records Open: Users have "unrestricted" access to open up to a maximum of 4 patient records at a time in the EHR
  Unrestricted, 2 record open: Users only opened 2 records at a time
- Unrestricted, 3 Records Open: Users have "unrestricted" access to open up to a maximum of 4 patient records at a time in the EHR
  Unrestricted, 1 record open: Users only opened 3 records at a time
- Unrestricted, 4 Records Open: Users have "unrestricted" access to open up to a maximum of 4 patient records at a time in the EHR
  Unrestricted, 4 records open: Users opened up to 4 records at a time
Arm/Group | Unrestricted, 1 Record Open | Unrestricted, 2 Records Open | Unrestricted, 3 Records Open | Unrestricted, 4 Records Open
Number analyzed (Participants) | 1687 | 1687 | 1687 | 1687
Number analyzed (Order sessions) | 1523585 | 303080 | 168387 | 267697
wrong order sessions / 100,000 sessions | 52.0 | 132.0 | 165.7 | 184.5
Statistical Analysis 1: Comparison: Unrestricted, 1 Record Open vs Unrestricted, 4 Records Open; Test type: Superiority; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: 19-month study period. The time frame for each participant varied.
Arm/Group | Unrestricted | Restricted
All-Cause Mortality (participants affected / at risk) | 0/1687 | 0/1669
Serious Adverse Events (participants affected / at risk) | 0/1687 | 0/1669
Other Adverse Events (participants affected / at risk) | 0/1687 | 0/1669

LIMITATIONS AND CAVEATS:
The outcome measure (Wrong-patient RAR measure) captures only one type of wrong-patient error; the study was conducted in a single health system and EHR platform, and therefore results may not be generalizable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/88/NCT02876588/Prot_SAP_000.pdf